CLINICAL TRIAL: NCT05806047
Title: Phase II Clinical Study of Combination of Chidamide and Fulvestrant for HR+/HER2- Breast Cancer That Has Failed Prior Adjuvant Therapy With CDK4/6 Inhibitors
Brief Title: Combination of Chidamide and Fulvestrant for HR+/HER2- Breast Cancer That Has Failed Previous CDK4/6 i Adjuvant Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C41
Record Dates: First submitted 2023-03-14; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Hormone Receptor-positive Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: chidamide combined with fulvestrant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide combined with fulvestrant (Experimental): chidamide combined with fulvestrant
  Interventions: Drug: chidamide combined with fulvestrant

INTERVENTIONS:
Drug: chidamide combined with fulvestrant — chidamide combined with fulvestrant

SUMMARY:
This trial is a single-arm study. The purpose of the trial is to evaluate the efficacy and safety of chidamide and fulvestrant in HR+/HER2- breast cancer that has failed prior adjuvant endocrine therapy with CDK4/6 inhibitors.

DETAILED DESCRIPTION:
The study was a single-center, single-arm, open trial design. Twenty-three patients with advanced HR+/HER2- breast cancer who had failed previous adjuvant treatment with CDK4/6 inhibitors in combination with endocrine therapy were treated with fulvestrant and chidamide.

ELIGIBILITY:
Inclusion Criteria:

1. Female, ≥18 years old;
2. ECOG score 0-1;
3. Predicted survival ≥3 months;
4. Patients with locally advanced and/or metastatic breast cancer confirmed by histopathology with positive ER expression and negative ER2 expression;
5. Patients who have relapsed or metastasized during or after CDK4/6 inhibitors combined with endocrine adjuvant therapy and have not received systemic antitumor therapy for the current stage of disease;
6. No previous treatment with fluvestran or use of fluvestran without proven treatment failure;
7. The time interval between non-endocrine therapy should be ≥2 weeks;
8. At least one extracranial measurable lesion as defined by RECIST V1.1 criteria;
9. The functions of vital organs meet the requirements;
10. Fertile subjects must have a negative pregnancy test 7 days before starting treatment and must use an appropriate contraceptive method during treatment and for three months after completion of treatment;
11. The patient is fully informed and voluntarily signs the informed consent.

Exclusion Criteria:

1. Prior treatment with any HDAC inhibitors;
2. Known allergy to the tested drug component;
3. inflammatory breast cancer at the time of screening;
4. pia meningeal metastasis confirmed by MRI or lumbar puncture;
5. Central nervous system metastasis confirmed by imaging;
6. To the best of the investigator's judgment, symptomatic visceral disease or any disease load or none is considered optimal Endocrine therapy options are not suitable for endocrine therapy;
7. Inability or unwillingness to swallow medication or receive intramuscular injections;
8. Gastrointestinal insufficiency or gastrointestinal disease (if not controlled) that may significantly affect study drug absorption Ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small intestine resection, etc.;
9. Patients with ascites, pleural effusion and pericardial effusion accompanied by clinical symptoms in the baseline period need drainage, or use it for the first time Patients with serous cavity drainage within 4 weeks before medication;
10. A history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency conditions, Or have a history of organ transplantation;
11. Other malignancies (cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and Thyroid cancer is excluded);
12. had undergone major surgical procedures or significant trauma within 4 weeks prior to the start of treatment, or was expected to undergo major surgery Surgical treatment;
13. Concomitant diseases that, in the investigator's judgment, seriously endanger patient safety or interfere with patient completion of the study (e.g.

    Severe hypertension, diabetes, thyroid disease, co-active hepatitis B/C, and other activities Sexual infection);
14. Inability to understand or follow research instructions and requirements;
15. The researcher decides that it is not suitable to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
ORR | max 6 months
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)

SECONDARY OUTCOMES:
PFS | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 1 years)
  time to progressive disease (according to RECIST1.1)
CBR | max 6 months
  The percentage of subjects with CR+PR+SD and last more than 24 weeks in all of the participants.
DOR | max 6 months
  Duration of Overall Response.The date of the first assessed PR/CR (according to RECIST 1.1) to the date of the first assessed tumor progression (according to RECIST 1.1) or death from any cause.